CLINICAL TRIAL: NCT06008782
Title: HEARS-SLP: Providing Speech Language Pathologist-Delivered Hearing Health Care to Individuals With Cognitive Impairment
Brief Title: HEARS-SLP: Providing SLP-Delivered Hearing Health Care to Individuals With Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB00218068; K23AG059900 (NIH)
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss; Dementia; Cognitive Impairment
MeSH Terms: conditions — Hearing Loss; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental): immediate treatment
  Interventions: Device: HEARS-SLP device; Behavioral: HEARS-SLP program
- Delayed treatment (Placebo Comparator): 1 month delayed treatment
  Interventions: Device: HEARS-SLP device; Behavioral: HEARS-SLP program

INTERVENTIONS:
Device: HEARS-SLP device — Tailored fitting and programming of a personal sound amplifier. This will be accompanied by a component of aural rehabilitation.
Behavioral: HEARS-SLP program — Tailored aural rehabilitation for participant and communication partner

SUMMARY:
Building upon the HEARS audiologist-community health worker (CHW) model, this study intervention will be delivered by a speech-language pathologist (SLP). The primary objective of the study is to develop and test an affordable and accessible hearing rehabilitative intervention that will be delivered by a SLP to individuals with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 - 100 years old
* English-speaking
* Lives at home
* Diagnosis of probable Alzheimer's Disease or other related dementia according to the core clinical criteria outlined in the National Institute on Aging (NIA) and Alzheimer's Association Guidelines
* Availability of caregiver/study partner to participate in all study-related visits and who provides ≥8 hours of weekly oversight/care
* Speech frequency pure tone average (0.5- 4 kHz) >25 db in the better-hearing ear; adult onset hearing loss
* Stable (for 2 weeks or longer) dosing of medication (e.g. antidepressants, antipsychotics) for neuropsychiatric symptoms

Exclusion Criteria:

* Current self-reported use of hearing aid or amplification device
* Medical contraindication to use hearing aids ( e.g. draining ears)
* Inability to participate in the 1-month follow up

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Neuropsychiatric Symptoms as assessed by the Neuropsychiatric Inventory (NPI-Q) | Baseline and 1 month post-intervention (immediate group). 1 month post-baseline (Delayed Group)
  Scoring: Each of the 12 NPI-Q domains contains a survey question that reflects symptoms of that domain. Initial responses to each domain question are "Yes" or "No". If the response to the question is "No", the informant goes to the next question. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale and the associated impact of the symptom manifestations on them using a 5-point scale. The NPI-Q provides symptom Severity and Distress ratings for each symptom reported, and total Severity and Distress scores reflecting the sum of individual domain scores. Total NPI-Q severity score is the sum of individual symptom scores, ranges from 0 to 36.
  SEVERITY of the symptom (how it affects the patient):
  1. = Mild (noticeable, but not a significant change)
  2. = Moderate (significant, but not a dramatic change)
  3. = Severe

SECONDARY OUTCOMES:
Change from Baseline in Health-related Quality of Life as assessed by the Quality of Life in Alzheimer's Disease (QOL-AD) scale | Baseline and 1 month post-intervention (immediate group). 1 month post-baseline (Delayed Group)
  Scoring for QOL-AD:
  Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.
  The total score is the sum of all 13 items. Total scores range from 13 to 52.
Change From Baseline in Hearing Specific Quality of life as assessed by the Hearing Handicap Inventory for the Elderly (HHIE-S) | Baseline and 1 month post-intervention (immediate group). 1 month post-baseline (Delayed Group)
  Higher scores indicate increased hearing handicap.
  Scoring:
  0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap An increase in the score from baseline (a positive number) indicates a worsening in hearing handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Oh, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No